CLINICAL TRIAL: NCT07299968
Title: Evaluation of the Welch Allyn Connex Spot Monitor in Measuring Respiratory Rate in the Emergency Department: a Prospective Observational Study Protocol
Brief Title: Accuracy of the Welch Allyn ConnexSpot Monitor in Measuring Respiratory Rate in the Emergency Department
Status: Not yet recruiting | Type: Observational
Sponsor: Dr. Rapszky Gabriella Anna (Other)
Collaborators: Semmelweis University (Other)
Responsible Party: Sponsor-Investigator, Dr. Rapszky Gabriella Anna, subinvestigator (PhD student, resident), Semmelweis University
Organization: Semmelweis University (Other)
Other Study IDs: SOK-LEGZ25
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-10

CONDITIONS: Respiratory Rate; Breathing Rate
Keywords: respiratory rate; emergency department; Welch
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational study will evaluate the accuracy of the Welch Allyn Connex Spot Monitor equipped with a Masimo SpO₂ finger sensor in measuring respiratory rate in the emergency department. Respiratory rate is a key predictor of patient deterioration, yet it is frequently measured inaccurately when assessed manually. In this study, respiratory rate values obtained by the monitor will be compared against manual counts performed by trained observers (physicians). An additional analysis will compare respiratory rates measured by trained observers with those recorded by triage nurses during triage. A subgroup analysis will also investigate whether cardiac arrhythmias influence measurement accuracy.

The aim is to examine if respiratory rates measured by the Welch Allyn Connex Spot Monitor are comparable to those obtained by trained observers and triage nurses in the emergency department.

DETAILED DESCRIPTION:
Design: prospective observational method comparison study

ELIGIBILITY:
Inclusion Criteria:

- all patients aged ≥18 years.

Exclusion Criteria:

* patients receiving invasive or non-invasive respiratory support;
* patients with disorders causing involuntary movements;
* skin or digit abnormalities preventing proper application of the pulse oximeter;
* clinically unstable patients on arrival (requiring immediate transfer to the resuscitation area);
* patients with a left ventricular assist device (LVAD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted on patients admitted to the Emergency Department of Semmelweis University.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Agreement between respiratory rate values measured by the Welch Allyn Connex Spot Monitor and manual counts performed by trained observers (reference standard) | During the emergency department visit (single measurement per participant).
  Respiratory rate will be measured simultaneously using the Welch Allyn Connex Spot Monitor and by trained observers performing manual counting over 60 seconds. Agreement between the two methods will be assessed using the Intraclass Correlation Coefficient and Bland-Altman analysis to evaluate bias and limits of agreement.

SECONDARY OUTCOMES:
Agreement between respiratory rate values measured by trained observers and those recorded by triage nurses during triage | During the emergency department visit (single measurement per participant).
  Respiratory rate measurements recorded by triage nurses during triage will be compared with manual 60-second counts performed by trained observers. Agreement between the two methods will be evaluated using the Intraclass Correlation Coefficient and Bland-Altman analysis to assess bias and limits of agreement.
Agreement between respiratory rate values measured by the Welch Allyn Connex Spot Monitor and manual counts performed by trained observers in patients with ECG-confirmed arrhytmias | During the emergency department visit (single measurement per participant).
  Respiratory rate measurements recorded by triage nurses during triage will be compared with manual 60-second spot measurements performed by trained observers. Agreement between the two methods will be evaluated using the Intraclass Correlation Coefficient and Bland-Altman analysis to assess bias and limits of agreement.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Emergency Medicine, Semmelweis University, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Semler MW, Stover DG, Copland AP, Hong G, Johnson MJ, Kriss MS, Otepka H, Wang L, Christman BW, Rice TW. Flash mob research: a single-day, multicenter, resident-directed study of respiratory rate. Chest. 2013 Jun;143(6):1740-1744. doi: 10.1378/chest.12-1837. PMID 23197319
- [Background] Loots FJ, Dekker I, Wang RC, van Zanten AR, Hopstaken RM, Verheij TJ, Giesen P, Smits M. The accuracy and feasibility of respiratory rate measurements in acutely ill adult patients by GPs: a mixed-methods study. BJGP Open. 2022 Dec 20;6(4):BJGPO.2022.0029. doi: 10.3399/BJGPO.2022.0029. Print 2022 Dec. PMID 35944945
- [Background] Edmonds ZV, Mower WR, Lovato LM, Lomeli R. The reliability of vital sign measurements. Ann Emerg Med. 2002 Mar;39(3):233-7. doi: 10.1067/mem.2002.122017. PMID 11867974
- [Background] Badawy J, Nguyen OK, Clark C, Halm EA, Makam AN. Is everyone really breathing 20 times a minute? Assessing epidemiology and variation in recorded respiratory rate in hospitalised adults. BMJ Qual Saf. 2017 Oct;26(10):832-836. doi: 10.1136/bmjqs-2017-006671. Epub 2017 Jun 26. PMID 28652259
- [Background] Leuvan CH, Mitchell I. Missed opportunities? An observational study of vital sign measurements. Crit Care Resusc. 2008 Jun;10(2):111-15. PMID 18522524
- [Background] Churpek MM, Yuen TC, Park SY, Meltzer DO, Hall JB, Edelson DP. Derivation of a cardiac arrest prediction model using ward vital signs*. Crit Care Med. 2012 Jul;40(7):2102-8. doi: 10.1097/CCM.0b013e318250aa5a. PMID 22584764
- [Background] Goldhill DR, McNarry AF, Mandersloot G, McGinley A. A physiologically-based early warning score for ward patients: the association between score and outcome. Anaesthesia. 2005 Jun;60(6):547-53. doi: 10.1111/j.1365-2044.2005.04186.x. PMID 15918825
- [Background] Mochizuki K, Shintani R, Mori K, Sato T, Sakaguchi O, Takeshige K, Nitta K, Imamura H. Importance of respiratory rate for the prediction of clinical deterioration after emergency department discharge: a single-center, case-control study. Acute Med Surg. 2016 Nov 10;4(2):172-178. doi: 10.1002/ams2.252. eCollection 2017 Apr. PMID 29123857
- [Background] Goldhill DR, White SA, Sumner A. Physiological values and procedures in the 24 h before ICU admission from the ward. Anaesthesia. 1999 Jun;54(6):529-34. doi: 10.1046/j.1365-2044.1999.00837.x. PMID 10403864
- See also: Product page for the Welch Allyn Connex Spot Monitor — https://www.hillrom.com/en/products/connex-spot-monitor/